CLINICAL TRIAL: NCT06106698
Title: Washed Microbiota Transplantation for Clostridioides Difficile Infection: a Real World Research
Brief Title: Washed Microbiota Transplantation for Clostridioides Difficile Infection
Status: Recruiting | Type: Observational
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: WMT-RWS-CDI
Record Dates: First submitted 2023-10-12; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-07

CONDITIONS: Clostridioides Difficile Infection
Keywords: washed microbiota transplantation; Clostridioides Difficile Infection; Intestinal infection; Antibiotic-associated Diarrhea
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — fecal and blood samples before and after intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: WMT — Washed microbiota transplantation refers to the infusion of washed microbiota from healthy donor into patients' gastrointestinal tract. Participants will receive one dose of WMT for CDI. During follow-up, those who have non-response or CDI recurrence within 4-week post-WMT will receive rescue WMT.

SUMMARY:
This is a real-world study to explore the safety and the efficacy of washed microbiota transplantation （WMT） for patients with Clostridioides Difficile Infection （CDI）.

DETAILED DESCRIPTION:
At least 12 subjects who meet all the inclusion criteria but do not meet any exclusion criteria will be enrolled in this study. Data of demographic characteristics, intestinal symptoms, medicine treatment usage and clinical outcomes will be collected. After treatment, they will enter the follow-up period （at least for 4-week post-WMT）for safety and efficacy evaluation. Subjects with no response and recurrence will receive salvage therapy, and the extended follow-up period will be performed.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to enter the study:

1. At the time of informed consent, male or non-pregnant or non-lactating female.
2. The diagnostic criteria for C. difficile infection are met during screening:

   1. Medical records confirming CDI prior to screening (laboratory tests are positive for Clostridium difficile or its toxin): Clostridium difficile toxin test is positive (determined by EIisa test), or colonoscopy indicates pseudomembranous enteritis; Or Glutamate dehydrogenase positive, toxin negative, there are obvious causes and diarrhea.
   2. CDI-related diarrhea episodes, i.e., defecation ≥3 times/day for at least two consecutive days with unformed stools (Bristol score 6-7).
3. The subject or his/her legal representative gives informed consent, fully understands the purpose of the study, is able to communicate effectively with the investigator, and comprehends and complies with the requirements set forth in the study.

Exclusion Criteria:

Subjects meeting any of the following exclusion criteria must be excluded from the study:

1. Subjects with immune deficiencies (such as HIV infection, or neutrophils <0.5×109/L in absolute value, or lymphocytes <0.5×109/L, etc.), or on immunosuppressants, or on medium to high doses of steroid hormones (≥20g/d of prednisone or equal doses of steroid hormones).
2. There is rectal outlet obstruction (such as rectal mucosal prolapse) or significant intestinal stenosis assessed by the investigator and colonic transendoscopic enteral tubing cannot be performed.
3. Confirmed or clinically suspected infection with pathogenic microorganisms other than Clostridium difficile prior to screening.
4. Have had major abdominal surgery (other than laparoscopic gallbladder or appendectomy), previous partial or total colectomy, previous partial small intestinal resection, or previous gastroduodenal surgery within 6 months prior to screening.
5. At the time of screening, the subject or his/her legal representative refuses to take effective contraception within 3 months after the last treatment.
6. According to the judgment of the investigator, the subjects are not suitable to participate in this clinical study, or participation in this clinical study cannot guarantee the rights and interests of the subjects.

Ages: 3 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: National patients with CDI receiving WMT will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-22 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of treatment-related adverse events (AE) assessed by CTCAE, Version 5.0 | Four-week post-WMT
  The severity of AE was graded as mild (grade 1), moderate (grade 2), severe/disabling (grade 3), life threatening (grade 4), and death (grade 5). All AE were divided in definitely, probably and possibly related to treatment. The treatment-related AE we focused on included microbiota-related AEs (e.g., infection, diarrhea, abdominal pain, etc.) and route of delivery related AEs (e.g., nausea, vomiting, etc.).

SECONDARY OUTCOMES:
The complete response rate of CDI-related diarrhea | Four-week post-WMT，eight-week post-WMT
  The complete response of CDI-related diarrhea was defined as there was no diarrhea (1-2 times/day) for at least two consecutive days (normal stool characteristics (Bristol score ≤5) after treatment.
Recurrence rate of CDI-related diarrhea. | Four-week post-WMT，eight-week post-WMT
  Recurrence was defined as the CDI-related diarrhea reappeared, and the Clostridium difficile toxin test was positive after achieving complete response.
Rate of major disease progression in CDI. | One-week post-WMT，Two-week post-WMT
  Disease progression refers to the worsening of symptoms associated with CDI, including increased diarrhea, toxic megacolon, organ failure, the need for emergency colectomy, and even death.
The incidence of treatment-related adverse events (AE) assessed by CTCAE, Version 5.0 | Eight-week post-WMT，six-month-post-WMT
  The severity of AE was graded as mild (grade 1), moderate (grade 2), severe/disabling (grade 3), life threatening (grade 4), and death (grade 5). All AE were divided in definitely, probably and possibly related to treatment. The treatment-related AE we focused on included microbiota-related AEs (e.g., infection, diarrhea, abdominal pain, etc.) and route of delivery related AEs (e.g., nausea, vomiting, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Faming Zhang, Principal Investigator — The Second Hospital of Nanjing Medical University
Locations (1):
- The second affiliated hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Guh AY, Mu Y, Winston LG, Johnston H, Olson D, Farley MM, Wilson LE, Holzbauer SM, Phipps EC, Dumyati GK, Beldavs ZG, Kainer MA, Karlsson M, Gerding DN, McDonald LC; Emerging Infections Program Clostridioides difficile Infection Working Group. Trends in U.S. Burden of Clostridioides difficile Infection and Outcomes. N Engl J Med. 2020 Apr 2;382(14):1320-1330. doi: 10.1056/NEJMoa1910215. PMID 32242357
- [Result] Antharam VC, Li EC, Ishmael A, Sharma A, Mai V, Rand KH, Wang GP. Intestinal dysbiosis and depletion of butyrogenic bacteria in Clostridium difficile infection and nosocomial diarrhea. J Clin Microbiol. 2013 Sep;51(9):2884-92. doi: 10.1128/JCM.00845-13. Epub 2013 Jun 26. PMID 23804381
- [Result] Pike CM, Theriot CM. Mechanisms of Colonization Resistance Against Clostridioides difficile. J Infect Dis. 2021 Jun 16;223(12 Suppl 2):S194-S200. doi: 10.1093/infdis/jiaa408. PMID 33326565
- [Result] Kelly CR, Fischer M, Allegretti JR, LaPlante K, Stewart DB, Limketkai BN, Stollman NH. Correction to: ACG Clinical Guidelines: Prevention, Diagnosis, and Treatment of Clostridioides difficile Infections. Am J Gastroenterol. 2022 Feb 1;117(2):358. doi: 10.14309/ajg.0000000000001529. No abstract available. PMID 34658366
- [Result] Drekonja D, Reich J, Gezahegn S, Greer N, Shaukat A, MacDonald R, Rutks I, Wilt TJ. Fecal Microbiota Transplantation for Clostridium difficile Infection: A Systematic Review. Ann Intern Med. 2015 May 5;162(9):630-8. doi: 10.7326/M14-2693. PMID 25938992
- [Result] Ademe M. Benefits of fecal microbiota transplantation: A comprehensive review. J Infect Dev Ctries. 2020 Oct 31;14(10):1074-1080. doi: 10.3855/jidc.12780. PMID 33175698
- [Result] Cammarota G, Ianiro G, Kelly CR, Mullish BH, Allegretti JR, Kassam Z, Putignani L, Fischer M, Keller JJ, Costello SP, Sokol H, Kump P, Satokari R, Kahn SA, Kao D, Arkkila P, Kuijper EJ, Vehreschild MJG, Pintus C, Lopetuso L, Masucci L, Scaldaferri F, Terveer EM, Nieuwdorp M, Lopez-Sanroman A, Kupcinskas J, Hart A, Tilg H, Gasbarrini A. International consensus conference on stool banking for faecal microbiota transplantation in clinical practice. Gut. 2019 Dec;68(12):2111-2121. doi: 10.1136/gutjnl-2019-319548. Epub 2019 Sep 28. PMID 31563878
- [Result] Ng SC, Kamm MA, Yeoh YK, Chan PKS, Zuo T, Tang W, Sood A, Andoh A, Ohmiya N, Zhou Y, Ooi CJ, Mahachai V, Wu CY, Zhang F, Sugano K, Chan FKL. Scientific frontiers in faecal microbiota transplantation: joint document of Asia-Pacific Association of Gastroenterology (APAGE) and Asia-Pacific Society for Digestive Endoscopy (APSDE). Gut. 2020 Jan;69(1):83-91. doi: 10.1136/gutjnl-2019-319407. Epub 2019 Oct 14. PMID 31611298
- [Result] van Nood E, Vrieze A, Nieuwdorp M, Fuentes S, Zoetendal EG, de Vos WM, Visser CE, Kuijper EJ, Bartelsman JF, Tijssen JG, Speelman P, Dijkgraaf MG, Keller JJ. Duodenal infusion of donor feces for recurrent Clostridium difficile. N Engl J Med. 2013 Jan 31;368(5):407-15. doi: 10.1056/NEJMoa1205037. Epub 2013 Jan 16. PMID 23323867